CLINICAL TRIAL: NCT06713772
Title: A Randomised Controlled Trial To Evaluate The Skin Closure Time, Parents' Satisfaction, Post Operative Mental Health, Wound Cosmesis and Wound Complication Of Skin Closure Using Adhesive Glue, Adhesive Tape And Suture In Paediatric Surgery Patients
Brief Title: To Evaluate The Skin Closure Time, Parents' Satisfaction, Post Operative Mental Health, Wound Cosmesis and Wound Complication Of Skin Closure Using Adhesive Glue, Adhesive Tape And Suture In Paediatric Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FF-2024-290
Record Dates: First submitted 2024-08-12; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Skin Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Adhesive glue (Active Comparator): Dermabond Mini, 0.36ml, Ethicon Johnson and Johnson, Somerville, New Jersey, USA
  Interventions: Device: Dermabond Mini, 0.36ml, Ethicon Johnson and Johnson, Somerville, New Jersey, USA
- Group B - Adhesive tape (Active Comparator): Steri-StripsTM (3M, St. Paul, Minnesota, USA
  Interventions: Device: Steri-StripsTM (3M, St. Paul, Minnesota, USA
- Group C - Suture (Active Comparator): Monosyn, B.Braun, 118 Pfieffewiesen, Melsungen, Germany
  Interventions: Device: Monosyn, B.Braun, 118 Pfieffewiesen, Melsungen, Germany

INTERVENTIONS:
Device: Dermabond Mini, 0.36ml, Ethicon Johnson and Johnson, Somerville, New Jersey, USA — Dermabond Mini, 0.36ml, Ethicon Johnson and Johnson, Somerville, New Jersey, USA
  Arms: Group A - Adhesive glue
Device: Steri-StripsTM (3M, St. Paul, Minnesota, USA — Steri-StripsTM (3M, St. Paul, Minnesota, USA
  Arms: Group B - Adhesive tape
Device: Monosyn, B.Braun, 118 Pfieffewiesen, Melsungen, Germany — Monosyn, B.Braun, 118 Pfieffewiesen, Melsungen, Germany
  Arms: Group C - Suture

SUMMARY:
This study is a randomised controlled trial to evaluate the skin closure time, parents' satisfaction, post operative mental health, wound cosmesis and wound complication of skin closure using adhesive glue, adhesive tape and suture in paediatric surgery patients.

Primary objective is to compare skin closure time required by using adhesive glue, adhesive tape and suture. Secondary objectives are to compare parents' satisfaction, post operative mental health, wound cosmesis and wound complication of skin closure using adhesive glue, adhesive tape and suture in paediatric surgery patients.

This study will be conducted from 26th August 2024 to 31st May 2025. It will take place at Hospital Pakar Kanak-Kanak UKM (HPKK), involving paediatric surgery patients undergoing clean or clean contaminated surgeries.

The sample size calculated is 30 per group, a total of 90 patients for three groups. The sampling method used is simple random sampling method.

In group A, skin will be closed using adhesive glue (Dermabond Mini, 0.36ml, Ethicon Johnson and Johnson, Somerville, New Jersey, USA). Skin closure in group B will be done using adhesive tape (Steri-StripsTM (3M, St. Paul, Minnesota, USA). In group C, skin will be closed using suture (Monosyn, B.Braun, 118 Pfieffewiesen, Melsungen, Germany) 4/0.

DETAILED DESCRIPTION:
This study is a randomised controlled trial to evaluate the skin closure time, parents' satisfaction, post operative mental health, wound cosmesis and wound complication of skin closure using adhesive glue, adhesive tape and suture in paediatric surgery patients.

Primary objective is to compare skin closure time required by using adhesive glue, adhesive tape and suture. Secondary objectives are to compare parents' satisfaction, post operative mental health, wound cosmesis and wound complication of skin closure using adhesive glue, adhesive tape and suture in paediatric surgery patients.

This study will be conducted from 26th August 2024 to 31st May 2025. It will take place at Hospital Pakar Kanak-Kanak UKM (HPKK), involving paediatric surgery patients undergoing clean or clean contaminated surgeries. Inclusion criteria includes patients aged 18 years or less, clean and clean contaminated surgery, wound length of 1-10cm, surgical wound amenable to closure with the three skin closure techniques. Exclusion criteria includes scrotal or penile incision, contaminated or dirty wound, repeated surgical procedures at the surgical site, wound that is not amenable to primary closure with the three techniques, patient with known allergy to cyanoacrylate, patients receiving chemotherapy, immunosuppression, systemic corticosteroids, or with known malignancy.

The sample size calculated is 30 per group, a total of 90 patients for three groups. The sampling method used is simple random sampling method.

In group A, skin will be closed using adhesive glue (Dermabond Mini, 0.36ml, Ethicon Johnson and Johnson, Somerville, New Jersey, USA). Skin closure in group B will be done using adhesive tape (Steri-StripsTM (3M, St. Paul, Minnesota, USA). In group C, skin will be closed using suture (Monosyn, B.Braun, 118 Pfieffewiesen, Melsungen, Germany) 4/0.

Primary outcome, skin closure time will be measured using stopwatch and documented in unit minutes and seconds. It will include the time taken for dressing application, but will not include the time taken for subcutaneous layer closure.

Secondary outcomes, parents' satisfaction will be measured in three aspects - ease of wound care, parents' feeling regarding wound management and satisfaction on wound cosmesis. These will be measured using Likert's scale at day 7 and 1 month post operation. Patient's post operative mental health will be measured in two aspects, post operative pain and patient's fear towards wound management post operation. Post operative pain will be assessed daily from day 1 to day 7. Visual Analog Scale will be used for patients more than 7 years old, whereas FLACC Scale will be used for patients less than 7 years old. Patient's fear towards wound management post operation will be measured using Children's Fear Scale at day 0 and day 7 post operation. Cosmetic appearance of skin will be assessed by using the Vancouver Scar Scale on the day 7 and 1 month. Wound complication will be assessed using ASEPSIS Score on the day 7 and 1 month post operation.

Data will be analysed using IBM SPSS Statistics Version 29. All continuous data (wound cosmesis, wound complication, post operative pain) will be checked for normality distribution using histogram, bell shape curve, skewness and kurtosis. If it is normally distributed, it will be presented in mean and standard deviation and further analysed and compared among three groups using analysis of variance (ANOVA). If it is not normally distributed, it will be presented in median and IQR and further analysed using Kruskal-Wallis test. P value < 0.050 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or less
* clean and clean contaminated surgery
* wound length of 1-10cm
* surgical wound amenable to closure with the three skin closure techniques

Exclusion Criteria:

* scrotal or penile incision
* contaminated or dirty wound
* repeated surgical procedures at the surgical site
* wound that is not amenable to primary closure with the three techniques
* patient with known allergy to cyanoacrylate
* patients receiving chemotherapy, immunosuppression, systemic corticosteroids, or with known malignancy

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Skin closure time | Day 0
  Skin closure time will be measured using stopwatch and documented in unit minutes and seconds. It will include the time taken for dressing application, but will not include the time taken for subcutaneous layer closure

SECONDARY OUTCOMES:
Parents' satisfaction | Day 7 and 1 month post operation
  Parents' satisfaction will be measured in three aspects - ease of wound care, parents' feeling regarding wound management and satisfaction on wound cosmesis. These will be measured using Likert's scale at day 7 and 1 month post operation
Post operative mental health (Post operative pain) | Day 1 to day 7
  Patient's post operative mental health (Post operative pain) - will be assessed daily from day 1 to day 7. Visual Analog Scale will be used for patients more than 7 years old, whereas FLACC Scale will be used for patients less than 7 years old.
Post operative mental health (Patient's fear towards wound management post operation) | Day 0 and day 7
  Patient's post operative mental health (Patient's fear towards wound management post operation) - will be measured using Children's Fear Scale at day 0 and day 7 post operation
Wound cosmesis | Day 7 and 1 month post operation
  Cosmetic appearance of skin will be assessed by using the Vancouver Scar Scale on the day 7 and 1 month
Wound complication | Day 7 and 1 month post operation
  Wound complication will be assessed using ASEPSIS Score on the day 7 and 1 month post operation

CONTACTS AND LOCATIONS:
Overall Officials: Marjimin Binti Osman, Principal Investigator — HUKM
Locations (1):
- HUKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No